CLINICAL TRIAL: NCT07265193
Title: The Workplace-Based, Multicomponent Hypertension Management Program in Patients Aged 18-60 Years: A Randomized Controlled Trial
Brief Title: The Workplace-Based Hypertension Management Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Yan-Feng Zhou, School of Public Health, Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 82404393
Record Dates: First submitted 2025-11-19; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Hypertension
Keywords: Hypertension; workplace health; behavioral intervention; randomized controlled trial; Kailuan study
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Workplace Health Management (Active Comparator): Routine workplace health education and management according to current guidelines, including routine health education, standard hypertension counseling, and usual workplace health services.
  Interventions: Other: Routine workplace health education and management according to current guidelines.
- Workplace-based Multicomponent Hypertension Management Program (Experimental): Multicomponent strategies, including default scheduling of BP monitoring and counseling sessions, personalized reminders via workplace digital systems, social comparison feedback using anonymized peer data, small incentives and commitment devices.
  Interventions: Behavioral: Workplace-based Multicomponent Hypertension Management Program

INTERVENTIONS:
Behavioral: Workplace-based Multicomponent Hypertension Management Program — Multicomponent strategies, including default scheduling of BP monitoring and counseling sessions, personalized reminders via workplace digital systems, social comparison feedback using anonymized peer data, small incentives and commitment devices.
  Arms: Workplace-based Multicomponent Hypertension Management Program
Other: Routine workplace health education and management according to current guidelines. — Routine workplace health education and management according to current guidelines, including routine health education, standard hypertension counseling, and usual workplace health services.
  Arms: Standard Workplace Health Management

SUMMARY:
This study aims to evaluate the effectiveness of a workplace-based, multicomponent hypertension management program for newly diagnosed patients. Investigators will recruit 512 participants (256 pairs) from the Kailuan Study in Tangshan, China. Participants will be randomly assigned to receive a Workplace-based Multicomponent Hypertension Management Program or Standard Workplace Health Management. The primary objective is to assess improvements in blood pressure control and hypertension-related health behaviors.

DETAILED DESCRIPTION:
Hypertension is a major public health issue worldwide, and workplace settings represent a critical intervention opportunity for middle-aged populations. Nudge theory provides a cost-effective and behaviorally informed approach to promote sustainable health behaviors. This randomized controlled trial (RCT) will explore mechanisms of health behavior promotion, evaluate the effectiveness of a nudge-based workplace health management strategy, and contribute to evidence-based hypertension prevention and control in China.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-60 years
* Newly diagnosed hypertension (per 2024 Chinese hypertension guideline criteria)
* Employed in Kailuan Group workplace settings
* Able to provide informed consent

Exclusion Criteria:

* Severe cardiovascular or renal disease at baseline
* Psychiatric disorders affecting compliance
* Pregnant or lactating women
* Participation in other intervention trials

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 512 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in systolic and diastolic blood pressure | up to 12 months
  Change in systolic and diastolic blood pressure from baseline to 12 months

SECONDARY OUTCOMES:
Changes in hypertension-related health behaviors | up to 12 months
  Changes in hypertension-related health behaviors (dietary intake, physical activity, medication adherence) at 12 months
Change in body mass index (BMI) | up to 12 months
  Change in body mass index (BMI) at 12 months
Work productivity and quality of life scores | up to 12 months
  Work productivity and quality of life scores (e.g., the European Quality of Life-5 Dimensions) at 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Yan-Feng Zhou, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be available upon reasonable request after publication of main trial results.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-11-28): https://cdn.clinicaltrials.gov/large-docs/93/NCT07265193/Prot_SAP_000.pdf